CLINICAL TRIAL: NCT03107169
Title: Fecal Microbiota Transplant Versus Vancomycin for Treatment of Initial Clostridium Difficile Infection
Brief Title: Treatment of Initial Clostridium Difficile Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Adrián Camacho-Ortiz, Dr., Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IF14-005
Record Dates: First submitted 2017-03-21; First posted 2017-04-11 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation; Vancomycin; Glycopeptides

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were randomized by a closed envelope method in a 1: 1 ratio to either oral vancomycin (every 6 h for 10-14 days) or a FMT-FURM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vancomycin (Active Comparator): Patients in this arm received vancomycin 250mg every 6 hrs for 10-14 days
  Interventions: Drug: Vancomycin
- FMT-FURM (Experimental): Patients in this arm receive FMT-FURM
  Interventions: Other: FMT

INTERVENTIONS:
Other: FMT — Patients in the FMT group received FMT-FURM
  Other Names: fecal microbiota transplant
  Arms: FMT-FURM
Drug: Vancomycin — Patients in the vancomycin group received oral vancomycin (250 mg every 6 h for 10-14 days)
  Other Names: Glycopeptide
  Arms: Vancomycin

SUMMARY:
Investigators designed an open, two-arm study to compare oral vancomycin with a fecal microbiota transplant (FMT) from a fecal donor-unrelated donor mix (FURM) as treatments for the first Clostridium difficile infection (CDI) episode among hospitalized patients.

DETAILED DESCRIPTION:
Investigators designed an open, two-arm study to compare oral vancomycin with an FMT-FURM as treatments for the first Clostridium difficile infection (CDI) episode among hospitalized patients. From each patient, a fecal sample was obtained at days 0, 3, and 7 after treatment. Specimens are cultured to isolate C. difficile, and C. difficile are assessed for the presence of genes encoding enterotoxin (tcdB), cytotoxin (tcdA), the binary toxin A (cdtA), binary toxin B (cdtB), and deletions within the negative regulator of toxin A and B production (tcdC) by polymerase chain reaction (PCR). The minimum inhibitory concentrations (MICs) of ciprofloxacin, moxifloxacin, erythromycin, clindamycin, vancomycin, metronidazole, linezolid, fidaxomicin, and tetracycline against C. difficile are measured using the agar dilution method. Fecal samples and FMT-FURM are analyzed by 16 subunit ribosomal ribonucleic acid (16S rRNA) metagenomic sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CDI (first episode)
* Older than 18 years old

Exclusion Criteria:

* Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Decrease in number of evacuations | up to a 2 days
  The cure of CDI was measured

IPD SHARING:
Plan to Share IPD: No